CLINICAL TRIAL: NCT06019091
Title: Optimal Frequency Used in Transcutaneous Electrical Nerve Stimulation (TENS) for Treating Pelvic Pain in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Elise De, Principal Investigator, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6485
Record Dates: First submitted 2023-06-07; First posted 2023-08-31 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Chronic Pelvic Pain
Keywords: Chronic pelvic pain; Chronic primary pelvic pain syndrome; Posterior tibial nerve stimulation; Transcutaneous electrical nerve stimulation; Neuromodulation

STUDY DESIGN:
Intervention Model Description: The participants will be randomized into three groups of 25 participants each for a total of 75 participants. The randomization will occur in blocks so that if the investigators need to terminate the study early there will be an equal number of participants in each group. The size of the blocks will also be kept secret for allocation concealment purposes. The randomization will be stratified by gender so that there is an equal number of participants from each gender in each group, reducing potential for gender as a confounding variable. Group 1 will be the low frequency set at 20 Hz. Group 2 will be the medium frequency set at 50 Hz. Group 3 will be the high frequency set 100 Hz. There is no sham group in this study as it has previously been found that posterior tibial TENS is effective and lasting. As such, all participants will be treated as a matter of routine medical care for pelvic pain.
Who Masked: Participant
Masking Description: There will be single blinding. Study participants/caretakers will not know which frequency has been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group 1, low frequency group, 20 Hz. (Active Comparator): Compass Health TENS 3000, 3 mode Analog Unit. Normal Mode (N), pulse width of 200 microseconds and an intensity to be determined in the office based upon when the participant feels sensitive to the TENS unit. Frequency (pulse rate) 20 Hz
  Interventions: Device: Compass Health TENS 3000, 3 mode Analog Unit
- Group 2, medium frequency, 50 Hz. (Active Comparator): Compass Health TENS 3000, 3 mode Analog Unit. Normal Mode (N), pulse width of 200 microseconds and an intensity to be determined in the office based upon when the participant feels sensitive to the TENS unit. Frequency (pulse rate) 50 Hz
  Interventions: Device: Compass Health TENS 3000, 3 mode Analog Unit
- Group 3, high frequency, 100 Hz. (Active Comparator): Compass Health TENS 3000, 3 mode Analog Unit. Normal Mode (N), a pulse width of 200 microseconds and an intensity to be determined in the office based upon when the participant feels sensitive to the TENS unit. Frequency (pulse rate) 100 Hz
  Interventions: Device: Compass Health TENS 3000, 3 mode Analog Unit

INTERVENTIONS:
Device: Compass Health TENS 3000, 3 mode Analog Unit — The TENS unit Compass Health TENS 3000, 3 mode Analog Unit will be configured based on randomization to 20 Hz, 50 Hz, or 100 Hz. Pulse width 200 microseconds, Normal (N) Mode. It will be used on the posterior tibial nerve via a patch that is supplied each day for 30 minutes of the day. These 30 minutes of intervention will occur at the participants most painful time of the day for their pain.

SUMMARY:
TENS (transcutaneous electrical nerve stimulation) is accepted as a standard treatment for chronic pelvic pain, but the best settings to recommend, including frequency of stimulation, have not been defined to date. This study aims to find the optimal frequency, also known as cycles per second or Hertz (Hz) for treating chronic pelvic pain using non-invasive skin-level electrical nerve stimulation. The investigators will see how people respond to (20Hz, 50Hz or 100Hz). The study will have a two week control period (one week that looks back retrospectively at the week prior and another week looking prospectively at the patient symptoms) with no TENS unit and the participants normal standard of care treatments. This will be followed by 2 weeks of active TENS treatment for 30 minutes a day at the most painful time of day for the participant. The participant will also be allowed to extend their trial to study for durability for up to 3 additional months after the initial study. Participants will be asked to fill out a VAS (visual analog scale), GUPI (genitourinary pain index) and TENS usage log weekly.

DETAILED DESCRIPTION:
Adults ages 18-90 years old who have first been given the standard of care therapy according to the AUA/EUA guidelines depending on their specific pain modality, first line treatments based on suspected etiology (for example pelvic floor physical therapy for high tone pelvic floor muscle dysfunction or amitriptyline for interstitial cystitis) without success will be defined as refractory. Participants who have plateaued on their response to current intervention strategies will be offered the TENS unit as an adjunct.

Participation will be offered by mail or in person. If by mail, the investigators will send the consent with the letter and questionnaires asking participants to call or bring the material if they would like to enroll. If the investigators speak to the subject over the phone, the investigators will discuss the study as comprehensively as if they were in the clinic. This will include explaining the concept of the TENS unit, the study itself, and clarifying any questions the participant has. Subsequently if they are interested in the study, the investigators will ask them to sign the consent and return it to us via mail or email.

Those whose pain symptomatology is above a threshold and who choose TENS therapy will be included in the study. The participants will be randomized into three groups of 25 participants each. The randomization will occur in blocks so that if the investigators need to terminate the study early there will be an equal number of participants in each group. The size of the blocks will also be kept secret for allocation concealment purposes. The randomization will be stratified by gender so that there is an equal number of participants from each gender in each group, reducing potential for gender as a confounding variable. Group 1 will be the low frequency set at 20 Hz. Group 2 will be the medium frequency set at 50 Hz. Group 3 will be the high frequency set 100 Hz. There is no sham group in this study as it has previously been found that posterior tibial TENS is effective and lasting. As such, all participants will be treated as a matter of routine medical care for pelvic pain. The investigators will use a fixed pulse width of 200 microseconds (uS), with continuous rather than biphasic stimulation. The investigators will aim to recruit 25 participants per group for a total of 75 participants.

Study Procedures

Screening Day 7/ Week 1 (in clinic or virtual): The first data points (Day 0) will take place in the clinic during the participant's routine visit or at the time of the participant's phone call seeking participation. If during a phone call seeking participation, this will be considered a study phone call, not a billable visit. The participant will fill out the VAS and GUPI. The participants will be taught how to fill out the pain assessment questionnaires (the VAS and GUPI, validated tools for measuring genitourinary pain and symptoms respectively). This can be done via paper to be brought into the office at their next checkup or via an emailed link through Qualtrics and uploaded to a spreadsheet in a protected AMC OneDrive. The baseline pain logs will be reviewed for sufficient severity of pain episodes and the participant will be randomized into the study if their pain is above the designated threshold: participants who record a pain scale of 4 or higher on any of the VAS scores or QOL score of 3 or higher on the GUPI question #9 will be eligible for the TENS study.

The GUPI and VAS will be collected at this time; this will record the participant's pain 1 week prior to the study and will be considered Day 7/week 1. The week 1 of screening will be combined with the first week of baseline measurement (week 2) for a 2-week lead-in. Participants will be taught how to complete a usage log (stating if the TENS was used each day and for how long in minutes) and will be asked to repeat this weekly. Participants will complete an inventory (the Treatment Map) of treatments tried prior to the TENS, throughout the study, and at the end.

Baseline Day 14/ Week 2: If the participant enrolls, they will be asked to continue logging pain (VAS and GUPI, on paper or via Qualtrics) for one week, with the week 1 screening and the week 2 baseline week totaling a 14-day control period. The control period will represent data (2 weeks of VAS and GUPI) with only baseline treatments and no TENS unit.

At week 2 (the end of the 2-week baseline, in person), participants will hand in scores and be randomized to a frequency. They will be given a TENS unit and taught how to use the unit. Teaching will include positioning of electrodes, as well as what buttons they are allowed to manipulate. The TENS unit settings will be pre-determined at the clinic and measures will be taken to ensure that the settings cannot be altered at home. The participant will be instructed not to open the TENS unit during the 2 treatment weeks of the study to ensure the settings are maintained. They will be instructed to continue only their baseline treatments.

Settings: The TENS unit used is a Compass Health TENS 3000, 3 mode Analog Unit. The participants' TENS unit will be set at Normal Mode (N), a pulse width of 200 microseconds and an intensity to be determined in the office based upon when the participant feels sensitive to the TENS unit. Frequency (pulse rate) will be determined by randomization. The participant will place the electrodes along the posterior tibial nerve on the medial ankle with a ground on the inner arch, each day for 30 minutes for a total of 14 days at the time of day typically associated with the worst pain or at the first opportunity for rest after this time.

Group 1 will be the low frequency group. This means that the TENS therapy will use a frequency of 20 Hz.

Group 2 will be the medium frequency group. This means that the TENS therapy will use a frequency of 50 Hz.

Group 3 will be the high frequency group. This means that the TENS therapy will use a frequency of 100 Hz.

Participants will be provided the TENS unit, its manual, and enough patches to last the 2 weeks of the treatment period. Participants will be given a weekly usage log, weekly pain VAS and weekly GUPI questionnaire logs again for 2 weeks they are actively using the TENS, with the option of paper or Qualtrics. In this log, the rating of pain by VAS and GUPI, the rating of genitourinary symptoms by GUPI, duration of TENS therapy, usage for every day of the week and adverse reactions to the TENS unit (rash) will be recorded.

Participants may be called during the 14-day treatment period to keep on track, address any concerns, questions, or any adverse reactions to TENS therapy by the physician or research staff. Their phone numbers will be maintained in the master key associated with the deidentified database in the AMC Onedrive protected research file for this purpose.

At 7 days and the end of the 14-day treatment period the visit can be performed either virtually or in the office. The 7-day visit will be considered purely a study visit and the 14 day visit a standard of care visit.

The completed week 3 and 4 VAS and GUPI, treatment usage documents will be returned. The participants will also be asked the question "Will you continue using TENS therapy for your pelvic pain?" Any persistent issues will be addressed during these visits as well and further options discussed.

For those who would like to continue the TENS unit, participants will be taught how to adjust settings and sites at home. Participants will be given repeat VAS and GUPI at 1, 2, and 3 months post-initial phase and seen again at 3 months as part of standard care. Here the investigators will review logs of what frequency patterns they developed with TENS usage on their own, if any. In this time participants may increase or decrease the frequency of their device anywhere in the range of 2 Hz to 150 Hz to see which they prefer most in this part of the trial. Participants will also be allowed to adjust pulse width (30 to 260 uS), mode (B N M), time (continuous, 15, 30 minutes), and intensity (1 to 8, 10-80mA) as desired. The only requests will be that they remove the device if any discomfort occurs and that they log their settings versus their response.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting with chronic pelvic pain (chronic/persistent pain that has been continuous or recurrent for at least three months (in accordance with EAU Guidelines).
2. Unsuccessful initial interventions based on initial assessments
3. Ability to provide informed consent and complete study requirements
4. Ability to complete a comprehensive history (including with an interpreter)

Exclusion Criteria:

1. Participants who have previously tried a new pharmacologic treatment for pelvic pain, neuromodulation or other alternative therapy for urologic disorders within the past 30 days
2. Inability to work a TENS unit
3. Any contraindications to usage of a TENS unit (pacemaker or other implantable device, lymphedema, pregnancy, malignancy, bleeding or clotting disorders, unhealthy tissue, seizure disorders, impaired cognition)
4. Any history of electrophysiologic heart disease or complications
5. Source of pain being an obvious anatomic issue requiring alternative treatment - for example urethral diverticulum, distal ureteric stone.
6. Participant who is pregnant
7. Participant with adhesive allergy either reported by the participant or upon chart review

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-04-18 (Estimated); Study Completion 2024-04-18 (Estimated)

PRIMARY OUTCOMES:
Percent change in VAS and GUPI pain questionnaires from baseline to after two weeks of therapy. | Three weeks
  The primary objective of the study is to compare the three TENS treatment groups after two weeks of active treatment, with respect to:
  The change in VAS and GUPI pain questionnaires from baseline to after two weeks of therapy.

SECONDARY OUTCOMES:
VAS questionnaire score comparison across the three TENS treatment groups | Three Weeks
  This secondary objective includes comparison of the three treatment groups with respect to the rating of VAS (Visual Analog Scale)scores separately (minimum value 0 least painful, maximum value 10 most painful). Analysis will be carried out to determine if there are time-dependent changes in questionnaire scores across the three TENS treatment groups.
  Pairwise comparisons of TENS groups will also be carried out to compare each arm with one another using Tukey's multiple comparison tests.
Time dependent changes in VAS questionnaire scores across the three TENS treatment groups | Three Weeks
  This secondary objective includes comparison of the three treatment groups with respect to the rating of VAS (Visual Analog Scale) scores overtime (by weekly diary entries) (minimum value 0 least pain, maximum value 10 most painful). Analysis will be carried out to determine if there are time-dependent changes in questionnaire scores across the three TENS treatment groups.
  Pairwise comparisons of TENS groups will also be carried out to compare each arm with one another using Tukey's multiple comparison tests.
GUPI questionnaire score comparison across the three TENS treatment groups | Three Weeks
  This secondary objective includes comparison of the three treatment groups with respect to the rating of GUPI (genitourinary pain index) scores separately (minimum value 0 delighted, maximum value 6 terrible). Analysis will be carried out to determine if there are time-dependent changes in questionnaire scores across the three TENS treatment groups.
  Pairwise comparisons of TENS groups will also be carried out to compare each arm with one another using Tukey's multiple comparison tests.
Time dependent changes in GUPI questionnaire scores across the three TENS treatment groups | Three Weeks
  This secondary objective includes comparison of the three treatment groups with respect to the rating of GUPI (genitourinary pain index) scores over time (minimum value 0 delighted, maximum value 6 terrible). Analysis will be carried out to determine if there are time-dependent changes in questionnaire scores across the three TENS treatment groups.
  Pairwise comparisons of TENS groups will also be carried out to compare each arm with one another using Tukey's multiple comparison tests.
Durability in optional extension phase of study | Three Months
  The investigators will again collect data at 1,2, and 3-months post-trial, asking how much the TENS has been used, to assess durability. This will be in a form that contains space to put the date and amount of time that the TENS unit was used for.

CONTACTS AND LOCATIONS:
Overall Officials: Elise De, MD, Principal Investigator — Urologist at Albany Medical Center
Locations (1):
- Albany Medical Center, Albany, New York, United States

REFERENCES:
- [Background] Sharma N, Rekha K, Srinivasan JK. Efficacy of transcutaneous electrical nerve stimulation in the treatment of chronic pelvic pain. J Midlife Health. 2017 Jan-Mar;8(1):36-39. doi: 10.4103/jmh.JMH_60_16. PMID 28458478
- [Background] Erol B, Danacioglu YO, Peters KM. Current advances in neuromodulation techniques in urology practices: A review of literature. Turk J Urol. 2021 Sep;47(5):375-385. doi: 10.5152/tud.2021.21152. PMID 35118977
- [Background] Cottrell AM, Schneider MP, Goonewardene S, Yuan Y, Baranowski AP, Engeler DS, Borovicka J, Dinis-Oliveira P, Elneil S, Hughes J, Messelink BJ, de C Williams AC. Benefits and Harms of Electrical Neuromodulation for Chronic Pelvic Pain: A Systematic Review. Eur Urol Focus. 2020 May 15;6(3):559-571. doi: 10.1016/j.euf.2019.09.011. Epub 2019 Oct 19. PMID 31636030
- [Background] Fall M, Baranowski AP, Elneil S, Engeler D, Hughes J, Messelink EJ, Oberpenning F, de C Williams AC; European Association of Urology. EAU guidelines on chronic pelvic pain. Eur Urol. 2010 Jan;57(1):35-48. doi: 10.1016/j.eururo.2009.08.020. Epub 2009 Aug 31. PMID 19733958
- [Background] Maher CF, Carey MP, Dwyer PL, Schluter PL. Percutaneous sacral nerve root neuromodulation for intractable interstitial cystitis. J Urol. 2001 Mar;165(3):884-6. PMID 11176493
- [Background] Tutolo M, Ammirati E, Heesakkers J, Kessler TM, Peters KM, Rashid T, Sievert KD, Spinelli M, Novara G, Van der Aa F, De Ridder D. Efficacy and Safety of Sacral and Percutaneous Tibial Neuromodulation in Non-neurogenic Lower Urinary Tract Dysfunction and Chronic Pelvic Pain: A Systematic Review of the Literature. Eur Urol. 2018 Mar;73(3):406-418. doi: 10.1016/j.eururo.2017.11.002. Epub 2018 Jan 12. PMID 29336927
- [Background] Tugay N, Akbayrak T, Demirturk F, Karakaya IC, Kocaacar O, Tugay U, Karakaya MG, Demirturk F. Effectiveness of transcutaneous electrical nerve stimulation and interferential current in primary dysmenorrhea. Pain Med. 2007 May-Jun;8(4):295-300. doi: 10.1111/j.1526-4637.2007.00308.x. PMID 17610451
- [Background] Mira TA, Giraldo PC, Yela DA, Benetti-Pinto CL. Effectiveness of complementary pain treatment for women with deep endometriosis through Transcutaneous Electrical Nerve Stimulation (TENS): randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2015 Nov;194:1-6. doi: 10.1016/j.ejogrb.2015.07.009. Epub 2015 Aug 6. PMID 26319650 (Retraction: PMID 30449593 Eur J Obstet Gynecol Reprod Biol. 2018 Nov 16;:)
- [Background] Johnson MI, Paley CA, Jones G, Mulvey MR, Wittkopf PG. Efficacy and safety of transcutaneous electrical nerve stimulation (TENS) for acute and chronic pain in adults: a systematic review and meta-analysis of 381 studies (the meta-TENS study). BMJ Open. 2022 Feb 10;12(2):e051073. doi: 10.1136/bmjopen-2021-051073. PMID 35144946
- [Background] Chen YJ, Zhou GY, Jin JH. [Transcutaneous electrical acupoint stimulation combined with auricular acupoint sticking for treatment of primary nocturnal enuresis]. Zhongguo Zhen Jiu. 2010 May;30(5):371-4. Chinese. PMID 20518171
- [Background] Tai C, Shen B, Chen M, Wang J, Liu H, Roppolo JR, de Groat WC. Suppression of bladder overactivity by activation of somatic afferent nerves in the foot. BJU Int. 2011 Jan;107(2):303-9. doi: 10.1111/j.1464-410X.2010.09358.x. PMID 20394612
- [Background] Vance CG, Rakel BA, Blodgett NP, DeSantana JM, Amendola A, Zimmerman MB, Walsh DM, Sluka KA. Effects of transcutaneous electrical nerve stimulation on pain, pain sensitivity, and function in people with knee osteoarthritis: a randomized controlled trial. Phys Ther. 2012 Jul;92(7):898-910. doi: 10.2522/ptj.20110183. Epub 2012 Mar 30. PMID 22466027
- [Background] Barroso U Jr, Viterbo W, Bittencourt J, Farias T, Lordelo P. Posterior tibial nerve stimulation vs parasacral transcutaneous neuromodulation for overactive bladder in children. J Urol. 2013 Aug;190(2):673-7. doi: 10.1016/j.juro.2013.02.034. Epub 2013 Feb 16. PMID 23422257

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT06019091/Prot_SAP_000.pdf